CLINICAL TRIAL: NCT07331103
Title: RESOLving INflammation Through Diet for Health Multicenter, Prospective Randomized, Controlled and Open- Label to Examine the Impact of a Diet Enriched in Omega 3 Fatty Acids of Animal and Vegetal Origin on Circulating Lipid-driven Pro-/Antiinflammatory Balance in Subjects at Moderate to High Cardiovascular Risk.
Brief Title: RESOLving INflammation Through Diet for Health (RESOLVIN)
Acronym: RESOLving
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mario Negri Institute for Pharmacological Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HORIZON-HLTH-2022-STAYHLTH-02; HORIZON-HLTH-2022- STAYHLTH-02 (Other Grant/Funding Number: CARE-IN HEALTH)
Record Dates: First submitted 2025-12-12; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Cardiovascualr Disease; Lipids; Inflammation; n-3 Polyunsatured Fatty Acids (n-3 PUFA)
Keywords: ASCVD; n-3 polyunsatured fatty acids; lipid driven/regulated vascular inflammation; n-3 PUFA; DHA; EPA; ALA
MeSH Terms: conditions — Inflammation | interventions — Fish Oils; Vitamin E

STUDY DESIGN:
Intervention Model Description: Multicenter, prospective randomized, controlled and open- label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Fish oil (Active Comparator): A total daily volume of 23.19 mL/day of fish oil.
  Interventions: Dietary Supplement: Fish Oil
- Camelina Sativa Oil (Active Comparator): a total volume of 30 mL/day + Vitamin E 24 mg.
  Interventions: Dietary Supplement: Camelina oil
- Control (Active Comparator): regular non-enriched diet + Vitamin E 24 mg
  Interventions: Dietary Supplement: Vitamin E

INTERVENTIONS:
Dietary Supplement: Fish Oil — 2262.5 mg DHA plus 1739.1 mh EPA
  Arms: Fish oil
Dietary Supplement: Camelina oil — 10g/day of ALA for a total volume of 30 mL/day
  Arms: Camelina Sativa Oil
Dietary Supplement: Vitamin E — a dose of 24 mg for the control group
  Arms: Control

SUMMARY:
Hyperlipidemia is the main driver of atherosclerotic cardiovascular disease (ASCVD), both through direct effects and as trigger of the chronic inflammation behind a cardiovascular health-to-disease transition. While lipid-lowering is an effective way to reduce the ASCVD risk, the residual risk remains high. In addition, a substantial proportion of ASCVD events occur in the absence of overt hyperlipidemia. Several lines of evidence ranging from experimental models to population studies and interventional clinical trials support chronic inflammation as the causal residual risk of CVD. The CVD risk-associated lipid classes contain fatty acids that can be liberated and metabolized into both inflammation-promoting as well as inflammation-resolving drivers, providing the rationale for focusing on this balance in the present project. Above all, the omega-3 fatty acid class can resolve inflammation but the potential impact is currently largely underestimated in CVD preventive recommendations. As cardiovascular preventive measures ease the burden placed on the individual, population, and on the health care system, it is critical to raise public awareness for chronic inflammation as a causative and modifiable cardiovascular risk factor and to provide tools for how to control and monitor it. As an alternative to marine sources, principally eicosapentaenoic acid (EPA) and less docosahexaenoic acid (DHA) can be endogenously produced from alpha-linolenic acid (ALA) found in plant oils. Secondarily the possibility to increase the consumption of vegetable oil may possibly decrease the environmental impacts of an intensive fishing and consecutive marine system imbalance. The overarching objective of CARE-IN-HEALTH is to assess if PUFAs may contribute to the resolution of the chronic lipid-driven/-regulated vascular inflammation in order to develop and test, in a real-life setting, tools for use in health care and by citizens to stay healthy by an adequate resolution of the chronic inflammation. The primary objective of the present study is to compare the effect on a lipid/inflammation-derived risk score of diets supplemented with polyunsaturated fatty acids (PUFA) of animal or vegetal origin with a nonenriched diet. The secondary objectives are a) to assess the acceptance of supplementation of diet with animal-derived or plant-derived PUFAs; b) to improve circulating lipid, inflammatory glycemic profile based on serial measurements of circulating biomarkers by means of PUFA supplementation. The study aims to identify a blueprint for how to control lipid-driven chronic inflammation by simple dietary interventions. Study population Participants to be considered for eligibility in the trial are adults aged >55 y, of both sexes (>=40% women), at moderate to high cardiovascular risk. The inclusion criteria are: Eligible participants will be at moderate to high SCORE2, SCORE2-OP and SCORE2-Diabetes risk level.

Non-eligible subjects will be those with:

* cardiovascular disease,
* established atherosclerotic vascular disease involving the coronary, peripheral, carotid, or aortic territories (identified by computerized tomography (CT) of coronary arteries, MRI, carotid or peripheral ultrasound imaging),
* chronic treatment with n-3 PUFA containing products (i.e., Vazkepa) or fibrates,
* a condition that interferes with the possibility to follow the dietary intervention, such as fish allergy or being a vegan,
* significant liver dysfunction,
* participation in another intervention clinical study. Participants will be centrally randomized by a web-based system to one of the 3 diets: 1) supplementation with 4 grams n-3 PUFAs (containing 2262.5 mg DHA plus 1739.1 mg EPA), 2) diet enriched with n-3 PUFAs of vegetable origin (Camelina Sativa Oil) + vitamin E 24 mg, and 3) regular uncontrolled diet + vitamin E 24 mg. The daily intake of 10 grams of ALA for participants randomized to Camelina Sativa Oil is equivalent to approximately 1500 mg of n-3 PUFAs. Fish oil and Camelina Sativa oil will be administered as liquid oils for the duration of 12 weeks. The addition of vitamin E is aimed at supplementing the same amount of this vitamin to participants. Eligible participants will undergo a clinical visit when also a blood sample will be taken at baseline and at 12 weeks follow-up. The main analysis will be performed according to a per protocol approach, therefore only participants compliant with study treatments will be included in the analysis. Primary objective: to compare the effect on a lipid/inflammation-derived risk score, based on circulating molecules, of diets enriched with PUFA of animal or vegetal origin with a non-enriched diet. Secondary objectives: a) to assess the acceptance of supplementation of diet with animal-derived or plant-derived PUFAs; b) to improve circulating lipidic/glycemic inflammatory profile. All 324 participants enrolled in the trial will have blood samples taken twice (at baseline and 12 weeks),

DETAILED DESCRIPTION:
This study aims to identify a blueprint for how to control lipid-driven chronic inflammation as well as tools to support the deployment of innovative personalized prevention of ASCVD by simple, easy dietary changes. In particular the primary endpoint is to compare the effect on a lipid/inflammation-derived risk score, of diets with supplementation of PUFA of animal or of vegetal origin with a non-enriched diet.

The secondary end points are: a) to assess the acceptance of supplementation of diet with animalderived or plant-derived PUFAs; b) to improve, by means of PUFA dietary supplementation, circulating lipidic/glycemic inflammatory profile based on serial measurements of circulating biomarkers. All subjects meeting inclusion/exclusion criteria will be centrally randomized by a web-based system to one of the three interventions:

1) supplementation with 4 grams of fish oil (containing 2262.5 mg DHA plus 1739.1 mg EPA, although a 10% variability due to the natural origin of the product must be considered), 2) diet enriched with 10 grams ALA of vegetable origin (Camelina Sativa Oil) + Vitamin E 24 mg, 3) regular non-enriched diet + Vitamin E 24 mg. Participants in RESOLVIN study will receive study agents from enrolment until 12 weeks follow-up.

The daily intake of EPA will be 1739 mg in participants assigned to fish oil, approximately 1500 mg for those assigned to 30 ml of camelina oil. The daily volume of camelina oil cannot be increased further without jeopardizing participant's compliance. The addition of vitamin E is aimed at supplementing the same amount of this vitamin to participants. The differential supplementation with vitamin E is requested by the different content of the vitamin in fish oil vs camelina oil. Both the fish oil and the camelina oil will be administered before food ingestion.

The study oils are ready to be ingested. Storage and dispensing of the study products will be done by the site pharmacists or by the responsible physician. The study oil ingestion will begin at randomization and will continue for 12 weeks. The addition of vitamin E is aimed at supplementing the same amount of this vitamin to participants assigned to camelina oil and controls. Vitamin E will be administered as solution, corresponding approx. to a daily dose of 24 mg.

At baseline, a blood sample for fatty acid analysis will be taken, demographic, clinical and treatment data will be collected, heart rate and blood pressure and waist circumference will be measured. At 12 weeks follow-up, clinical information about tolerance of diets enriched by PUFAs and any clinical event will be collected. Heart rate, blood pressure and waist circumference will be measured; blood will be sampled at baseline and 12 weeks to be processed stored and then shipped to the central biobank. All participants will be asking to complete a 15-item dietary assessment questionnaire at baseline and 12 weeks follow-up. Central randomization will be performed in a 1:1:1 ratio. The following information will be required:

* center/GP code, participant initials, date of birth, sex.
* inclusion and exclusion criteria.
* signed and dated informed consent. A participant will be considered randomized when the randomization system will assign the participants identification number according to a pre-established randomization list. Randomization will be stratified by Centre/GP.

ELIGIBILITY:
Inclusion Criteria:

* Participants are subjects >55 y old from both sexes (>=40% women) with moderate to high cardiovascular risk (ANNEX 1: SCORE2, SCORE2-OP and SCORE2-Diabetes assessment).

Exclusion Criteria:

* cardiovascular disease,
* established atherosclerotic vascular disease involving the coronary, peripheral, carotid, or aortic territories (identified by computerized tomography (CT) of coronary arteries, MRI, carotid or peripheral ultrasound imaging),
* chronic treatment with n-3 PUFA containing products (i.e., Vazkepa),
* a condition that interferes with the possibility to follow the dietary intervention, such as fish allergy or being a vegan,
* significant liver dysfunction,
* participation in another intervention clinical study.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 324 (Estimated)
Dates: Start 2025-11-26 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
the effect on a lipidomic/inflammation- derived risk score based on plasma biomarkers | up to 12 weeks
  to compare the effect on a lipid/inflammation-derived risk scoremoderate= 50-69 years: 5 to 10%; >70 years: 7.5 to <15%; high=50-69 years: >10%; 70 years >15%), based on circulating molecules, of diets enriched with PUFA of animal or vegetal origin with a non-enriched diet.
Primary objective | 18 months
  The primary endpoint is to compare the effect on a lipidomic/inflammation-derived risk score based on plasma biomarkers, of diets with supplementation with PUFA of animal or vegetal origin with a non-enriched diet.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Meessen, phD, Principal Investigator — Laboratory Clinical Research in Brain and Cardiovascular Injury Istituto di Ricerche Farmacologiche Mario Negri IRCCS
Locations (5):
- Italy (5):
  - Dr. Antonella Todesca, Avellino, AV
  - Dr. Tommaso Reginato, Arese, MI
  - Istituto di Ricerche Farmacologiche Mario Negri, Milan, MI
  - Dr. Giosafatte Zappia, Paderno Dugnano, MI
  - Ospedale Madonna delle Grazie Matera, Matera, MT

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dietary supplementation with n-3 polyunsaturated fatty acids and vitamin E after myocardial infarction: results of the GISSI-Prevenzione trial. Gruppo Italiano per lo Studio della Sopravvivenza nell'Infarto miocardico. Lancet. 1999 Aug 7;354(9177):447-55. PMID 10465168
- [Background] Ridker PM, Everett BM, Thuren T, MacFadyen JG, Chang WH, Ballantyne C, Fonseca F, Nicolau J, Koenig W, Anker SD, Kastelein JJP, Cornel JH, Pais P, Pella D, Genest J, Cifkova R, Lorenzatti A, Forster T, Kobalava Z, Vida-Simiti L, Flather M, Shimokawa H, Ogawa H, Dellborg M, Rossi PRF, Troquay RPT, Libby P, Glynn RJ; CANTOS Trial Group. Antiinflammatory Therapy with Canakinumab for Atherosclerotic Disease. N Engl J Med. 2017 Sep 21;377(12):1119-1131. doi: 10.1056/NEJMoa1707914. Epub 2017 Aug 27. PMID 28845751
- [Background] Tunon J, Badimon L, Bochaton-Piallat ML, Cariou B, Daemen MJ, Egido J, Evans PC, Hoefer IE, Ketelhuth DFJ, Lutgens E, Matter CM, Monaco C, Steffens S, Stroes E, Vindis C, Weber C, Back M. Identifying the anti-inflammatory response to lipid lowering therapy: a position paper from the working group on atherosclerosis and vascular biology of the European Society of Cardiology. Cardiovasc Res. 2019 Jan 1;115(1):10-19. doi: 10.1093/cvr/cvy293. PMID 30534957
- [Background] Visseren FLJ, Mach F, Smulders YM, Carballo D, Koskinas KC, Back M, Benetos A, Biffi A, Boavida JM, Capodanno D, Cosyns B, Crawford C, Davos CH, Desormais I, Di Angelantonio E, Franco OH, Halvorsen S, Hobbs FDR, Hollander M, Jankowska EA, Michal M, Sacco S, Sattar N, Tokgozoglu L, Tonstad S, Tsioufis KP, van Dis I, van Gelder IC, Wanner C, Williams B; ESC National Cardiac Societies; ESC Scientific Document Group. 2021 ESC Guidelines on cardiovascular disease prevention in clinical practice. Eur Heart J. 2021 Sep 7;42(34):3227-3337. doi: 10.1093/eurheartj/ehab484. No abstract available. PMID 34458905
- [Background] Back M, Yurdagul A Jr, Tabas I, Oorni K, Kovanen PT. Inflammation and its resolution in atherosclerosis: mediators and therapeutic opportunities. Nat Rev Cardiol. 2019 Jul;16(7):389-406. doi: 10.1038/s41569-019-0169-2. PMID 30846875